CLINICAL TRIAL: NCT07124078
Title: A Phase 2, Randomized, Open-Label Study of Axatilimab Versus Best Available Therapy in Pediatric Participants With Chronic Graft-Versus-Host Disease After at Least 2 Prior Lines of Systemic Therapy (AGAVE-256)
Brief Title: A Study to Evaluate Axatilimab Versus Best Available Therapy in Pediatric Participants With Chronic Graft-Versus-Host Disease After at Least 2 Prior Lines of Systemic Therapy (AGAVE-256)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA034176-256
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; Calcineurin Inhibitors; Cyclosporine; Tacrolimus; Photopheresis; Mycophenolic Acid; Everolimus; Sirolimus; Rituximab; Imatinib Mesylate; Methotrexate; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axatilimab (Experimental): Axatilimab at the protocol-defined dose.
  Interventions: Drug: INCA034176
- Best available Treatment (BAT) (Experimental): Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Interventions: Drug: Best available Treatment (BAT)

INTERVENTIONS:
Drug: INCA034176 — Axatilimab at the protocol-defined dose.
  Other Names: Axatilimab
  Arms: Axatilimab
Drug: Best available Treatment (BAT) — Best Available Therapy (BAT) will be selected by the Investigator for each participant. BAT may not include experimental agents (i.e. those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements.
  Other Names: BAT could include:; • Calcineurin inhibitor (cyclosporine or tacrolimus); • Extracorporeal photopheresis (ECP); • Mycophenolate mofetil (MMF); • A mammalian target of rapamycin (mTOR) inhibitor (everolimus or sirolimus); • Rituximab; • Imatinib; • Methotrexate; • Ibrutinib
  Arms: Best available Treatment (BAT)

SUMMARY:
This study will be conducted to compare Axatilimab Versus Best Available Therapy in Pediatric Participants With Chronic Graft Versus Host Disease After at Least 2 Prior Lines of Systemic Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 2 to < 18 years at the time of signing the informed consent.
* Active, moderate to severe cGVHD, requiring systemic immune suppression.
* Participants with refractory or recurrent cGVHD who have received at least 2 lines of systemic therapy, including corticosteroids and ruxolitinib.
* Concomitant use of systemic corticosteroids is allowed. Participants on systemic corticosteroids must be on a stable dose of corticosteroids for at least 2 weeks prior to C1D1. Topical and inhaled corticosteroid agents are allowed.
* Participants must accept to be treated with one of the following BAT options on C1D1: CNI (cyclosporine or tacrolimus), ECP, MMF, an mTOR inhibitor (everolimus or sirolimus), rituximab, imatinib, methotrexate, or ibrutinib.
* History of allo-HCT from any donor HLA type (related or unrelated donor with any degree of HLA matching) using any graft source (bone marrow, peripheral blood stem cells, or cord blood). Recipients of myeloablative, nonmyeloablative, or reduced-intensity conditioning are eligible.

Exclusion Criteria:

* Receipt of more than 1 prior allo-HCT. Prior autologous HCT is allowed.
* Evidence of relapse of hematologic disease or treatment for relapse after the allo-SCT was performed, including DLI for the treatment of molecular relapse. Note: Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible.
* Systemic treatment with CNIs or mTOR inhibitors started within 2 weeks prior to C1D1.
* Severe renal impairment, that is, GFR < 30 mL/min/1.73 m2 as estimated using modified Schwartz formula, or end-stage renal disease on dialysis.
* Impaired liver function, defined as total bilirubin > 1.5 × ULN and/or ALT and AST > 3 × ULN in participants with no evidence of liver cGVHD.
* History of acute or chronic pancreatitis.
* Active, symptomatic myositis.
* Female adolescent participants who are pregnant or breastfeeding.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response (OR) at 6 months | 6 months
  Defined for each treatment group as complete response (CR) or partial response (PR) at 6 months (Cycle 7 Day 1, 28-day cycles) in the absence of new systemic therapy for cGVHD. Responses defined by the 2014 NIH consensus criteria.

SECONDARY OUTCOMES:
Pharmacokinetics Parameter (PK): Cmax of axatilimab | Up to 5 years
  Defined as maximum observed plasma concentration of axatilimab.
Pharmacokinetics Parameter: Tmax of axatilimab | Up to 5 years
  Defined as the time to reach the maximum plasma concentration of axatilimab.
Pharmacokinetics Parameter: Cmin of axatilimab | Up to 5 years
  Defined as the minimum observed plasma concentration of axatilimab.
Pharmacokinetics Parameter: AUC(0-t) of axatilimab | Up to 5 years
  Defined as the area under the concentration-time curve up to the last measurable concentration of axatilimab.
Pharmacokinetics Parameter: AUC 0-∞ of axatilimab | Up to 5 years
  Defined as the area under the concentration-time curve from 0 to infinity of axatilimab.
Pharmacokinetics Parameter: CL of axatilimab | Up to 5 years
  Defined as the apparent oral dose clearance of axatilimab.
Pharmacokinetics Parameter: Vz of axatilimab | Up to 5 years
  Defined as the apparent oral dose volume of distribution of axatilimab.
Pharmacokinetics Parameter: t1/2 of axatilimab | Up to 5 years
  Defined as the apparent terminal phase disposition half-life of axatilimab.
Best Overall Response (BOR) | Up to 5 years
  Defined as best response of CR or PR in the first 6 months (up to and including Cycle 7 Day 1), and at any timepoint up to the initiation of new systemic therapy for cGVHD.
Overall Response at 12 months | 12 months
  Defined as CR or PR at 12 months in the absence of new systemic therapy for cGVHD.
Duration of Response (DOR) (in responders only) | Up to 5 years
  Defined as the time from the date of first response (PR or CR) to the date of progression of cGVHD, initiation of new systemic treatment for cGVHD, or death from any cause, whichever comes first. An additional measure of response durability will consider DOR as the time from the date of first response to the date of new systemic therapy for cGVHD or death from any cause, whichever occurs first.
Organ-specific response | Up to 5 years
  Organ-specific response as defined in the protocol.
Percent reduction in daily corticosteroid dose at 6 months | 6 months
  Defined as Percent reduction in daily corticosteroid dose at Cycle 7 Day 1, and participants successfully tapered off all corticosteroids at Cycle 7 Day 1.
Changes in parameters collected using the pediatric stem cell quality of life (Q0L) questionnaire (PedsQL Stem Cell Transplant Module) | Up to 5 years
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 5 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (39):
- United States (9):
  - City of Hope Medical Center, Duarte, California
  - Lucile Packard Child Hospital End, Stanford, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Adventhealth Pediatric Cellular Therapy and Blood and Marrow Transplant, Orlando, Florida
  - Emory Childrens Center, Atlanta, Georgia
  - Memorial Sloan Kettering, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (2):
  - Hôpital Universitaire Des Enfants Reine Fabiola, Brussels
  - Universite Catholique de Louvain (Ucl) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Germany (7):
  - Charite Campus Virchow, Berlin
  - Klinikum Der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main
  - Universitaetsklinikum Freiburg Zentrum Fuer Kinderheilkunde Und Jugendmedizin Klinik Iv, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover (Mhh) - Zentrum Fuer Kinderheilkunde Und Jugendmedizin - Klinik Fue, Hanover
  - Universitaeres Krebszentrum Leipzig (Uccl)-Universitatsklinikum Leipzig Aor, Leipzig
  - University Hospital Regensburg, Regensburg
- Italy (6):
  - Irccs - Aou Di Bologna - Sant'Orsola Malpighi, Bologna
  - Irccs Istituto G. Gaslini, Universita Di Genova, Genova
  - Fondazione Irccs San Gerardo Dei Tintori, Monza
  - Azienda Ospedaliera Universitaria Di Padova, Padua
  - Fondazione Irccs Policlinico San Matteo Di Pavia Oncoematologia Pediatrica, Universita Di Pavia, Pavia
  - Irccs Ospedale Pediatrico Bambino Gesu, Rome
- Spain (5):
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga- Hospital Materno Infantil, Málaga
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Universitat de Valencia - Hospital Universitari I Politecnic La Fe de Valencia, Valencia
- United Kingdom (10):
  - Birmingham Children'S Hospital - Birmingham Women'S and Children'S Nhs Foundation Trust, Birmingham
  - Addenbrooke'S Hospital - Cambridge University Hospitals Nhs Foundation Trust, Cambridge
  - The Royal Hospital For Children - Glasgow Health Board, Glasgow
  - Leeds Childrens Hospital, Leeds
  - University College London Hospitals - University College London Hospitals Nhs Foundation Trust, London
  - St Mary'S Hospital, Paddington - Imperial College Healthcare Nhs Trust, London
  - Great Ormond Street Hospital For Children Nhs Foundation Trust, London
  - Royal Manchester Children'S Hospital - Manchester University Nhs Foundation Trust, Manchester
  - Royal Victoria Infirmary - the Newcastle Upon Tyne Hospitals Nhs Foundation Trust, Newcastle
  - Sheffield Children'S Hospital - Sheffield Children'S Nhs Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate Axatilimab Versus Best Available Therapy in Pediatric Participants With Chronic Graft-Versus-Host Disease After at Least 2 Prior Lines of Systemic Therapy (AGAVE-256) — https://incyteclinicaltrials.com/studies/inca034176-256